CLINICAL TRIAL: NCT03679013
Title: A Pilot Study Comparing the Effectiveness of an Opioid- Sparing Analgesic Regimen and an Opioid Based Regimen on Post- Operative Pain Control in Cardiac Surgery Patients (INOVA OPIOID
Brief Title: Effectiveness of an Opioid Sparing Pain Regimen in Cardiac Surgery
Acronym: INOVAOPIOID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Ramesh Singh, Cardiothoracic Surgeon, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-3002
Record Dates: First submitted 2018-09-05; First posted 2018-09-20 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
Keywords: cardiac; surgery; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid based standard of care regimen. (Other): Inova Heart and Vascular Institute (IHVI) opioid based standard of care regimen given for post operative cardiac surgery pain.
  Interventions: Drug: Opiate based pain regimen.
- Opioid sparing pain regimen. (Experimental): Multimodal pain regimen consisting of PO Gabapentin paired with intravenous Acetaminophen given for post operative cardiac surgery pain.
  Interventions: Drug: Oral Gabapentin and Intravenous Acetaminophen (IV APAP)

INTERVENTIONS:
Drug: Oral Gabapentin and Intravenous Acetaminophen (IV APAP) — Scheduled multimodal pain regimen consisting of oral Gabapentin paired with intravenous Acetaminophen following cardiopulmonary bypass surgery.
  Other Names: PO Gabapentin and IV APAP
  Arms: Opioid sparing pain regimen.
Drug: Opiate based pain regimen. — Standard of care opiate based pain regimen.
  Other Names: Post operative opioids
  Arms: Opioid based standard of care regimen.

SUMMARY:
The Inova Heart and Vascular Institute (IHVI) perform over 300 coronary artery bypass graft (CABG) surgeries per year. While opioid medications are the institutional standard of care for post-operative pain therapy little is known about the variation in pain scores, incidence of post- operative complications, and cost of hospitalization when an alternative multimodal pain regimen consisting of oral Gabapentin and intravenous Acetaminophen (IV APAP) is utilized.

The objective is to determine whether there is a substantial difference in pain scores, incidence of post-operative complications, and costs associated with hospitalization when a non-opioid multimodal pain regimen is utilized A single- center, open label, prospective, randomized, controlled clinical trial comprised of 20 total patients who have undergone isolated CABG at the IHVI will be conducted. Separate cohorts will include patients receiving opioid medications post-operatively (Group 1) and patients receiving the non-opioid regimen of oral Gabapentin and IV APAP (Group 2) to be followed for 72 hours post CABG surgery.

Main outcome measures include pain scores in both study groups, requests for breakthrough pain medication in both groups, gastrointestinal and respiratory complications of ileus and reduction in tidal volumes or forced vital capacity (FVC) at baseline and at 72 hours,increase in serum AST/ALT, and comparison of cost of hospitalization between groups.

The objective of this pilot study is to provide evidence that multimodal pain therapy utilizing IV APAP and PO Gabapentin will provide more effective pain relief than standard of care opioids as evidenced by pain scores <2. And the reduced consumption of opioids will lead to a reduction in ileus, no increase in AST/ALT, post-operative tidal volumes as assessed by incentive spirometry comparable to pre- surgical values, while also showing a positive effect on the cost of hospitalization.

DETAILED DESCRIPTION:
The Cardiovascular Intensive Care Unit (CVICU) of the Inova Heart and Vascular Institute (IHVI) will be the setting of this clinical trial involving two groups of subjects and comparing the opiate based standard of care regimen currently adopted (Group 1) at the IHVI with a treatment group (Group 2). Group 2 will receive a scheduled multimodal pain regimen consisting of PO (pro ora [oral]) Gabapentin paired with intravenous Acetaminophen. Opioids will be available for breakthrough pain in the treatment group for pain scores greater than 4. The outcomes of total opioid consumption and minimum/ maximum pain scores will be assessed at the 24 hours, 48 hours, 72 hours, and PRN (pro re nata [as the situation demands]) timepoints. Assessment will include amount of opioids consumed in both groups as well as number of requests for breakthrough pain medication in Group 2.

Minimum and maximum pain scores in all study groups will be assessed via Numeric Rating Scale (0-10) as per Inova Health System (IHS) policy; 'Pain Management for the Adult Population', at 24 hours, 48 hours, 72 hours, and PRN with opioid requests in all groups and opioid administration follow up within one hour as per IHS inpatient medication administration policy. Follow up medication administration scores will not be recorded as part of study results.

Secondary assessments will include the incidence of ileus both during hospitalization, increase in aspartate aminotransferase (AST)/ alanine aminotransferase (ALT), post-operative tidal volumes as assessed by incentive spirometry as compared to pre- surgical values, time from Cardiovascular Intensive Care Unit (CVICU) arrival to extubation in both groups, and the effects of an opioid based regimen versus an opioid sparing regimen on cost of medication and hospitalization.

The investigators hypothesize that a scheduled opioid- sparing pain regimen consisting of intravenous Acetaminophen IV APAP and PO Gabapentin for 48 hours post- operatively will reduce opioid consumption while maintaining adequate pain relief as evidenced by pain scores less than two (2), and a reduction in opioid consumption, and that reduced opioid consumption will lead to a reduction in the incidence of ileus, an opioid related side effect, no increase in AST/ALT, post-operative tidal volumes as assessed by incentive spirometry comparable to pre- surgical values, and demonstrate a positive effect on the cost of medication and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 18 and 85 years old.
2. Elective or urgent surgery requiring sternotomy approach
3. Subject is able to read and has signed and dated the informed consent document including authorization permitting release of personal health information (PHI) approved by the Inova Institutional Review Board (IRB).

Exclusion Criteria:

1. Patients lacking enteral access on post-operative day 0
2. Inability to communicate
3. Active chronic pain with opioid therapy
4. Active chronic use of gabapentin or pregabalin
5. Active substance abuse
6. Current self- report of alcoholism
7. End stage renal disease
8. Active renal dialysis therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Singh, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Heart and Vascular institute, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen.
Started | 8 | 11
Completed | 8 | 7
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen. | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Full Range); unit: years] | 68.1 [62.8 to 73.4] | 65.5 [57.7 to 73.3] | 66.8 [57.7 to 73.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 8 | 9 | 17
  Race: African American | 0 | 0 | 0
  Race: Asian | 0 | 1 | 1
  Race: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Requests for Breakthrough Opioid Pain Medication in Opioid Standard of Care Regimen Compared to Non-opioid Multimodal Pain Relief Regimen (Experimental Group).
Description: Number of patients with requests for breakthrough pain medication. Requests for breakthrough pain medication is defined as having pain scores >4 using the Numeric Rating Scale: a dimensional measurement of pain intensity; 0-10 scale for scoring pain (0= "no pain", 10"worst pain imaginable")
Time Frame: 24 hours, 48 hours, 72 hours after post-surgical treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen.
Number analyzed (Participants) | 8 | 11
Participants
  24 hours | 7 | 2
  48 hours | 7 | 1
  72 hours | 1 | 1

2. Primary Outcome: Average Pain Score at 24, 48 and 72 Hours Post-operatively
Description: Participants were assessed by rating their pain according to the Numeric Rating Scale: a dimensional measurement of pain intensity; 0-10 scale for scoring pain (0= "no pain", 10="worst pain imaginable")
  The minimum and maximum pain scores per participant were aggregated at timepoints of 24 hours, 48 hours, and 72 hours after the start of post-operative treatment
Time Frame: at 24, 48, and 72 hours after the start of post-operative treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen.
Number analyzed (Participants) | 8 | 11
score on a scale
  Minimum Pain Score at 24 hours | 1 [0 to 3] | 0.09 [0 to 1]
  Maximum Pain Score at 24 hours | 7 [4 to 10] | 3.18 [0 to 5]
  Minimum Pain Score at 48 hours | 1 [0 to 3] | 0.18 [0 to 1]
  Maximum Pain Score at 48 hours | 6.75 [3 to 8] | 3.64 [0 to 6]
  Minimum Pain Score at 72 hours | 0 [0 to 0] | 0 [0 to 0]
  Maximum Pain Score at 72 hours | 2.5 [0 to 5] | 2.36 [0 to 6]

3. Secondary Outcome: Number of Participants With Ileus During Hospitalization
Description: The number of participants with occurrences of ileus during hospitalization.
Time Frame: Surgery completion through study completion up to one week.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen.
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: randomization through 72 hours after randomization
Arm/Group | Opioid Based Standard of Care Regimen. | Opioid Sparing Pain Regimen.
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03679013/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03679013/ICF_001.pdf